## **Study Title:**

Preventing Alcohol and Other Drug Use and Violence Among Latino Youth

**NCT #:** 

NCT05240313

## **Date of Document:**

January 2, 2022 (first drafted)
February 10, 2025 (edited for clinicaltrials.gov resubmission)

## **Statistical Analysis Plan**

We conducted a descriptive analysis of participant demographics and a basic description of baseline and follow-up outcomes. The goal of this study was to examine the feasibility and acceptability of the adapted intervention—data for this aim were based on retention and the qualitative assessment of participants and study facilitators.